CLINICAL TRIAL: NCT03827629
Title: A Phase 1, Open-Label, Randomized, Crossover, Comparative Bioavailability Study of Naloxone Nasal Spray and Naloxone Hydrochloride Intramuscular Injection in Healthy Volunteers
Brief Title: A Study to Compare Bioavailability of Naloxone Nasal Spray and Naloxone Hydrochloride (HCl) Intramuscular Injection (IM) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INS012-17-108
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: Treatment Sequence A-B-C (Experimental): Participants received Treatment A on Day 1 of Period 1, Treatment B on Day 1 of Period 2, and Treatment C on Day 1 of Period 3.
  Interventions: Drug: Treatment A: Naloxone Nasal Spray; Drug: Treatment B: Naloxone Nasal Spray; Drug: Treatment C: Naloxone HCL Intramuscular (IM) Injection
- Cohort 2: Treatment Sequence B-C-A (Experimental): Participants received Treatment B on Day 1 of Period 1, Treatment C on Day 1 of Period 2, and Treatment A on Day 1 of Period 3.
  Interventions: Drug: Treatment A: Naloxone Nasal Spray; Drug: Treatment B: Naloxone Nasal Spray; Drug: Treatment C: Naloxone HCL Intramuscular (IM) Injection
- Cohort 3: Treatment Sequence C-A-B (Experimental): Participants received Treatment C on Day 1 of Period 1, Treatment A on Day 1 of Period 2, and Treatment B on Day 1 of Period 3.
  Interventions: Drug: Treatment A: Naloxone Nasal Spray; Drug: Treatment B: Naloxone Nasal Spray; Drug: Treatment C: Naloxone HCL Intramuscular (IM) Injection
- Cohort 4: Treatment Sequence A-C-B (Experimental): Participants received Treatment A on Day 1 of Period 1, Treatment C on Day 1 of Period 2, and Treatment B on Day 1 of Period 3.
  Interventions: Drug: Treatment A: Naloxone Nasal Spray; Drug: Treatment B: Naloxone Nasal Spray; Drug: Treatment C: Naloxone HCL Intramuscular (IM) Injection
- Cohort 5: Treatment Sequence C-B-A (Experimental): Participants received Treatment C on Day 1 of Period 1, Treatment B on Day 1 of Period 2, and Treatment A on Day 1 of Period 3.
  Interventions: Drug: Treatment A: Naloxone Nasal Spray; Drug: Treatment B: Naloxone Nasal Spray; Drug: Treatment C: Naloxone HCL Intramuscular (IM) Injection
- Cohort 6: Treatment Sequence B-A-C (Experimental): Participants received Treatment B on Day 1 of Period 1, Treatment A on Day 1 of Period 2, and Treatment C on Day 1 of Period 3.
  Interventions: Drug: Treatment A: Naloxone Nasal Spray; Drug: Treatment B: Naloxone Nasal Spray; Drug: Treatment C: Naloxone HCL Intramuscular (IM) Injection

INTERVENTIONS:
Drug: Treatment A: Naloxone Nasal Spray — Participants received naloxone nasal spray following a 10 hour fast.
Drug: Treatment B: Naloxone Nasal Spray — Participants received naloxone nasal spray following a 10 hour fast.
Drug: Treatment C: Naloxone HCL Intramuscular (IM) Injection — Participants received naloxone HCl IM injection following a 10 hour fast.

SUMMARY:
The main objective of this study is to compare early exposures of two test formulations of Naloxone Nasal Spray with the reference formulation of Naloxone HCl IM Injection under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* A minimum body weight of 50 kg and a body mass index (BMI) between 18.0 and 32.0 kilogram per square meter (kg/m2)
* A seated blood pressure between 90 and 140 millimeters of mercury (mmHg) systolic/50 and 90 mmHg diastolic (inclusive)
* Female subjects had a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test at screening

Exclusion Criteria:

* A known allergy or history of significant adverse reaction to naloxone, other opioids or related compounds, or to any of the excipients.
* Any documented clinically significant infection, injury, or illness within 1 month prior to screening.
* An active malignancy of any type, or had been diagnosed with cancer within 5 years prior to screening.
* A documented history of alcohol or drug abuse/dependence/misuse or narcotic analgesic abuse/dependence/misuse within 2 years prior to screening. Alcohol abuse was defined as greater than 14 drinks per week.
* Positive serology test for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) at screening.
* A positive urine test result for alcohol, drugs, or cotinine at screening or check-in.
* A condition that the Investigator believed would have interfered with the ability to provide informed consent or comply with study instructions, or that could confound the interpretation of the study results or put the subject at undue risk.
* Used any opioids for 30 days prior to Day 1.
* Required treatment with monoamine oxidase inhibitors (MAOIs) within 30 days prior to Day 1 and during the study.
* Presence of an ongoing upper respiratory infection, rhinitis, rhinorrhea, or nasal congestion.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of Unconjugated Naloxone | Pre-dose and at multiple time points up to 1 hour post-dose
Partial Area Under the Concentration Curve (AUC) of Unconjugated Naloxone | Pre-dose and at multiple time points up to 1 hour post-dose

SECONDARY OUTCOMES:
Area Under the Curve from Time 0 to the Last Measured Concentration (AUC0-t) of Unconjugated Naloxone | Pre-dose and at multiple time points up to 24 hours post-dose
Area Under the Curve from Time 0 to Infinity (AUC0-inf) of Unconjugated Naloxone | Pre-dose and at multiple time points up to 24 hours post-dose
Percentage of AUC0-inf Obtained by Extrapolation (AUCextrap) of Unconjugated Naloxone | Pre-dose and at multiple time points up to 24 hours post-dose
Maximum Plasma Concentration (Cmax) of Unconjugated Naloxone | Pre-dose and at multiple time points up to 24 hours post-dose
Time to Reach Maximum Plasma Concentration (Tmax) of Unconjugated Naloxone | Pre-dose and at multiple time points up to 24 hours post-dose
Last Quantifiable Concentration (Clast) of Unconjugated Naloxone | Pre-dose and at multiple time points up to 24 hours post-dose
Time of the Last Quantifiable Concentration (Tlast) of Unconjugated Naloxone | Pre-dose and at multiple time points up to 24 hours post-dose
Time Prior to the First Measurable (Non-Zero) Concentration (Tlag) of Unconjugated Naloxone | Pre-dose and at multiple time points up to 24 hours post-dose
Elimination Rate Constant (λz) of Unconjugated Naloxone | Pre-dose and at multiple time points up to 24 hours post-dose
Elimination Half-Life (t1/2) of Unconjugated Naloxone | Pre-dose and at multiple time points up to 24 hours post-dose
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 10
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product during the course of a clinical investigation. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not thought to be related to the investigational product. A serious AE (SAE) is any AE that results in death, is life threatening, requires hospitalization or prolongs existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is medically significant or requires intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni DeCastro, Study Director — INSYS Therapeutics Inc
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States